CLINICAL TRIAL: NCT02603224
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single and Multiple Dose-Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Activity of MRG-201 Following Local Intradermal Injection in Normal Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetic Study of MRG-201 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: miRagen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRG201-30-001
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRG-201 (Experimental)
  Interventions: Drug: MRG-201
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MRG-201 — Intradermal injection of single ascending doses and multiple ascending doses in healthy volunteers.
  Arms: MRG-201
Drug: Placebo — Intradermal injection of placebo at a second site in healthy volunteers. Each subject will serve as their own control.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of the investigational drug, MRG-201, in healthy volunteers. MRG-201 is designed to mimic the activity of a molecule called miR-29 that decreases the expression of collagen and other proteins that are involved in scar formation. MRG-201 is being studied to determine if it can limit the formation of fibrous scar tissue in certain diseases.

MRG-201 will be tested in healthy volunteers by injection into intact skin or adjacent to a short skin incision. Volunteers may receive one or several doses of MRG-201, and will be monitored for local reactions in the skin, signs or symptoms of adverse effects on the body, and for the levels of MRG-201 in the blood over time. Skin biopsies will also be collected to study how cells in the skin respond when exposed to MRG-201.

DETAILED DESCRIPTION:
Study Design:

Cohorts of 3-6 healthy male volunteers, ages 18-45, will receive single or multiple ascending doses of MRG-201 by intradermal injection at one site and placebo at a second site over a period of up to 15 days, with follow-up for up to 28 days after the last dose to determine the maximum tolerated dose in intact or incised normal skin and the tendency for active drug to diffuse through the skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18 and 45 years of age inclusive
* Body Mass Index (BMI) 18-35 kg/m^2 inclusive
* Must have 2 regions on the lower back/upper buttocks free of striae, scars, tattoos or other skin pathologies
* If engaged in sexual relations with a female of child-bearing potential, must be willing to use two effective contraceptive methods throughout the treatment period and for at least 12 weeks after the last treatment administration

Exclusion Criteria:

* Clinically significant abnormalities in medical history or physical exam which in the opinion of the Investigator would make the subject unsuitable for inclusion in the study
* History of cutaneous disorder that could interfere with the study or put the subject at risk
* History of renal or liver dysfunction or evidence of renal or liver dysfunction at screening
* History of clinically significant anemia or evidence of clinically significant anemia at screening
* Positive for blood borne pathogen (HBV, HCV, HIV) at screening
* Prior malignancies within the past 3 years (allowing squamous cell and basal cell carcinomas that have been successfully treated)
* Use of systemic steroids or topical steroids on the target area within two months of the Baseline visit or use of topical steroids outside the target area within 14 days of the Baseline visit
* Use of an investigational small molecule drug within 28 days of the baseline visit or use of an investigational oligonucleotide or biologic drug within 90 days of the baseline visit

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MRG-201 based on vital signs, physical examination, clinical laboratory tests, ECG, and incidence and severity of adverse events | Up to 43 days

SECONDARY OUTCOMES:
Area under the plasma concentration vs. time curve (AUC) of MRG-201 following single and repeat doses | Up to 17 days
Peak plasma concentration (Cmax) of MRG-201 following single and repeat doses | Up to 17 days

OTHER OUTCOMES:
Exploratory assessment of the levels of miR-29 target mRNAs in skin following treatment with MRG-201 or placebo using the Nanostring nCounter® analysis system | Up to 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilad S. Gordon, MD, Study Director — miRagen Therapeutics, Inc.
Locations (1):
- Innovaderm Research, Inc., Montreal, Quebec, Canada